CLINICAL TRIAL: NCT05619445
Title: Feasibility of Egg-Based Diet Interventions and Assessing Perinatal Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Idaho (Other)
Collaborators: University of Nevada, Las Vegas (Other); University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-117
Record Dates: First submitted 2022-10-24; First posted 2022-11-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Depression; Anxiety; Stress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole Liquid Egg (Experimental): Whole Liquid Eggs
  Interventions: Other: Whole Liquid Egg
- Plant-Based Egg Substitute (Experimental): Plant-Based Egg Substitute
  Interventions: Other: Plant-based Egg Substitute

INTERVENTIONS:
Other: Whole Liquid Egg — Subjects will consume 2 fluid ounces of whole liquid eggs per day for 120 days.
  Arms: Whole Liquid Egg
Other: Plant-based Egg Substitute — Subjects will consume 2 fluid ounces of liquid plant-based egg substitute (JUST eggs) per day for 120 days.
  Arms: Plant-Based Egg Substitute

SUMMARY:
The goals of this study are to assess the feasibility and acceptability of a dietary intervention to increase choline intake through whole foods (eggs) in pregnant and lactating women for mental health benefits. We will achieve these goals through the following specific aims:

1. To determine the effects of including eggs as a source of choline in the diets of pregnant and lactating women on biomarkers, we will measure concentrations of choline and choline metabolites in maternal serum and breastmilk at 24-26 weeks gestation and 4-6 weeks postpartum.
2. To evaluate adherence to a food-based dietary choline intervention in pregnant and lactating women, we will track intake via daily photo and written food logs.
3. To assess the feasibility of collecting repeated measures of dietary intake and maternal depression, anxiety, and stress in the perinatal period, we will track completion rates for project surveys.

The data from this study will inform the design and sample size calculations for a longitudinal cohort study that will assess neurological outcomes for both mother and child and follow the offspring over time to reassess mental health and cognitive development in preschool-aged children.

Choline is an underconsumed nutrient of concern for public health, specifically during pregnancy and lactation. There is limited data on biomarker or health outcomes related to perinatal choline intake. Determining relationships between perinatal choline intake and maternal mental health has the potential to impact public health by ultimately informing development of nutrition education materials in the clinical setting focused on encouraging maternal perinatal choline intake through whole foods such as eggs.

DETAILED DESCRIPTION:
Subjects will be recruited from community sites, such as health clinics and recreation centers. Practitioners and recreation center directors will collaborate by sharing a recruitment flyer with patients and clients. Doctor's clearance is not required for participation, but potential subjects may discuss the study with their physician. Potential subjects will complete an online screening form. Eligible subjects (n=30) will be 18 to 26 weeks pregnant (at study start, mid-July), have access to internet and an electronic devise (phone, tablet, or computer), and be willing to consume eggs and consent to study participation. Eligible subjects will be sent an electronic informed consent and be contacted by study personnel. Study personnel will review the consent either in person, via phone, or via zoom. Those eligible for the study will be randomly assigned to the dietary intervention groups: whole liquid eggs (n=15) or plant-based liquid egg substitute (JUST Egg) (n=15).

After consenting, subjects will complete baseline surveys. Baseline survey data collected will include an online demographic and health history questionnaire, food frequency questionnaire, 24-hour dietary recall, and self-report surveys to assess depressive symptoms, anxiety, perceived stress, and perceived social support. Subjects will complete all assessments online (via Qualtrics) using their own electronic devices, including phone, tablet, or computer, from the comfort of their own home.

Subjects will then be scheduled to come to the Ramsay Research unit (RRU) for fasted blood draw (overnight fast, 8 hours). Subjects will be scheduled between 7:30am and 11am. The RRU is not a CLIA-certified laboratory. It is an approved research laboratory. Blood will be processed at the RRU and sent to the Chen lab on the UI Moscow campus for cortisol analysis and to the University of North Carolina Nutrition Research Institute for choline analysis. At this baseline visit, subjects will also receive the first 30 day supply of the assigned dietary intervention along with a simple recipe book to offer ideas for preparation in case subjects are not familiar with how to prepare liquid eggs and to reduce monotony and palate fatigue. Subjects will also receive a measuring cup and a diet log along with instructions for consuming the intervention food and reporting intake daily via photos and written log. Researchers will answer any questions. Subjects will receive baseline data collection compensation.

Subjects will pick up additional dietary intervention products at the Carmelita Spencer Foods laboratory every 30 days (total of 120 days). Alternatively, research personnel will deliver products to subjects' homes in the Moscow area.

Subjects will be asked to take a photo of each meal that incorporates their assigned dietary intervention food before and after eating. These photos will be sent to the study phone via text message and uploaded to the PI's secure university One Drive account.

Subjects will be asked to complete additional online 24-hour diet recalls at week 9-10 of the intervention (about week 35-36 gestation), and week 18-19 of the intervention (about 4-5 weeks postpartum).

At week 4-6 postpartum, subjects will complete a short survey online describing birth-related outcomes and experience and self-report surveys to assess depressive symptoms, anxiety, perceived stress, and perceived social support.

Also at 4-6 weeks postpartum, subjects will come to the Ramsay Research Unit for fasted blood draw (overnight fast, 8 hours) and to provide a sample of breastmilk. Subjects will be scheduled between 7:30am and 11am. Subjects will be asked to refrain from feeding their infant on one breast for the 2 hours prior to collection. An electronic breast pump will be provided and a lactation specialist will be available to assist in this collection. Subjects will be asked for a full expression from one breast. Blood will be processed as described above. Breastmilk will sent to the UNC Nutrition Research Institute for choline analysis.

This will complete the data collection and subjects will receive study completion compensation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 26 weeks pregnant
* have access to internet and an electronic device (phone, tablet, or computer)
* willing to consume eggs

Exclusion Criteria:

* score 11 or higher on the Edinburgh Postnatal Depression Scale
* under 19 years of age
* non-English speaking
* pregnant with multiples
* consume a vegan diet
* self-reported use of alcohol or drugs during pregnancy
* have diagnosed egg allergy
* have physical, cognitive, or logistical limitations to being able to follow the study protocol
* do not plan to breastfeed

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Serum Choline | Baseline
  Blood will be collected and analyzed via liquid chromatography-stable isotope dilution-multiple reaction monitoring mass spectrometry
Serum Choline | 4-6 weeks postpartum
  Blood will be collected and analyzed via liquid chromatography-stable isotope dilution-multiple reaction monitoring mass spectrometry
Adherence | Daily through the dietary intervention (120 days)
  Daily photo and written diet logs will be analyzed to determine dietary intake of the intervention foods
Feasibility/Compliance | Through study completion, approximately 4 months
  Percent of subjects who complete all study surveys will be calculated to report feasibility of collecting repeated measures of dietary intake and mental health surveys.

SECONDARY OUTCOMES:
Breastmilk Choline | 4-6 weeks postpartum
  Breastmilk will be collected and analyzed via liquid chromatography-stable isotope dilution-multiple reaction monitoring mass spectrometry
Depression | Baseline
  Maternal depressive symptoms will be measured via the Edinburgh Postnatal Depression Scale. Maximum score is 30. Higher scores indicate increased symptoms of depression.
Depression | 4-6 weeks postpartum
  Maternal depressive symptoms will be measured via the Edinburgh Postnatal Depression Scale. Maximum score is 30. Higher scores indicate increased symptoms of depression.
Anxiety | Baseline
  Maternal anxiety will be measured with the 31-item perinatal anxiety screening scale. Maximum score is 93. Higher scores indicate higher symptoms of anxiety.
Anxiety | 4-6 weeks postpartum
  Maternal anxiety will be measured with the 31-item perinatal anxiety screening scale. Maximum score is 93. Higher scores indicate higher symptoms of anxiety.
Stress | Baseline
  Maternal perceived stress levels will be characterized via the Perceived Stress Scale. The maximum score is 56. Higher scores indicate higher levels of perceived stress.
Stress | 4-6 weeks postpartum
  Maternal perceived stress levels will be characterized via the Perceived Stress Scale. The maximum score is 56. Higher scores indicate higher levels of perceived stress.
Perceived social support | Baseline
  Subjects will complete the Multidimensional Scale of Perceived Social Support. The maximum score is 7. Higher scores indicate higher levels of perceived support.
Perceived social support | 4-6 weeks postpartum
  Subjects will complete the Multidimensional Scale of Perceived Social Support. The maximum score is 7. Higher scores indicate higher levels of perceived support.
Serum cortisol | Baseline
  Blood draw will be analyzed for concentration of serum cortisol using an enzyme-linked immunosorbent assay
Serum cortisol | 4-6 weeks postpartum
  Blood draw will be analyzed for concentration of serum cortisol using an enzyme-linked immunosorbent assay

CONTACTS AND LOCATIONS:
Overall Officials: Annie J Roe, PhD, Principal Investigator — University of Idaho
Locations (1):
- University of Idaho, Moscow, Idaho, United States

IPD SHARING:
Plan to Share IPD: No